CLINICAL TRIAL: NCT02061917
Title: Switching From Usual Brand Cigarettes to a Tobacco-heating Cigarette or Snus - A Multi-center Evaluation of Health-related Quality of Life Assessments and Biomarkers of Exposure and Harm
Brief Title: Switching From Usual Brand Cigarettes to a Tobacco-heating Cigarette or Snus
Acronym: QoL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R.J. Reynolds Tobacco Company (Industry)
Collaborators: Analytisch-biologisches Forschungslabor GmbH (Industry); Arista Laboratories (Unknown); Covance (Industry); Covance IVRS (Unknown); Pacific Biomarkers (Other); University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSD-0702
Record Dates: First submitted 2014-02-05; First posted 2014-02-13 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Cigarette Smoking
Keywords: Biomarkers; Tobacco; Tobacco-heating; Smokeless Tobacco; Snus; Smoking; Exposure; Quality of Life
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use; Smoking | interventions — Tobacco, Smokeless

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tobacco-Heating Cigarette (Experimental): A group of 44 subjects who smoke and are switched to a tobacco-heating cigarette
  Interventions: Other: Tobacco-Heating Cigarette
- Snus (Smokeless Tobacco) (Experimental): A group of 43 subjects who smoke and are switched to snus (smokeless tobacco)
  Interventions: Other: Snus (Smokeless Tobacco)
- Tobacco-Burning Cigarette (Experimental): A group of 44 subjects who smoke and are switched to a tobacco-burning ultra-low machine yield cigarette
  Interventions: Other: Tobacco-Burning Cigarette

INTERVENTIONS:
Other: Tobacco-Heating Cigarette — Smokers switched to a tobacco-heating cigarette for 24 weeks
  Arms: Tobacco-Heating Cigarette
Other: Snus (Smokeless Tobacco) — Smokers switched to snus product for 24 weeks
  Arms: Snus (Smokeless Tobacco)
Other: Tobacco-Burning Cigarette — Smokers switched to a tobacco-burning cigarette for 24 weeks
  Arms: Tobacco-Burning Cigarette

SUMMARY:
To evaluate selected biomarkers of tobacco exposure and biomarkers of harm and assess quality of life measures in smokers randomly switched from their usual brand of cigarette to one of three test products: (1) a tobacco-heating cigarette; (2) snus (smokeless tobacco); or (3) an ultra-low machine yield tobacco-burning cigarette.

DETAILED DESCRIPTION:
A randomized, multi-center, 4-group study of health status measures and biomarkers in subjects who smoke and are switched to either a tobacco-heating cigarette, snus, or a tobacco-burning cigarette, with a non-treatment group of never-smokers.

Primary Objectives:

* Evaluate select biomarkers of tobacco exposure and biomarkers of harm from subjects who smoke and who are switched to a tobacco-heating cigarette, snus, or a tobacco-burning cigarette.
* Evaluate ability of a tobacco-heating cigarette and snus to modify patient-reported Chronic Obstructive Pulmonary Disease (COPD)-related health status in subjects who smoke and are switched to either a tobacco-heating cigarette or snus relative to a control group (a tobacco-burning ultra-low machine yield [ULMY]) cigarette.
* Assess subject compliance.

Secondary Objectives:

* Measure amount and repeatability of smoke components yielded from the cigarettes (yield in use) and determine relative uptake of selected smoke components.
* Evaluate the ability of a tobacco-heating cigarette and snus to modify general health status as measured by self-administered health questionnaires in subjects who smoke and are switched to either a tobacco-heating cigarette or snus relative to a control group (a tobacco-burning ULMY cigarette).
* Compare health status measures in smokers who are switched to a tobacco-heating cigarette to smokers who are switched to snus.
* Compare baseline data from all tobacco-using groups to baseline data from the never-smoking (non-treatment) group.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, between 28 and 55 years of age, inclusive.
* Cigarette-only smokers who currently smoked at least 15 cigarettes daily and who smoked for at least 10 years prior to Week 0 (i.e., chronic cigarette smokers).
* Smokers not intending to quit smoking, but willing to switch their tobacco product (intent to quit was defined as intending to make or making a quit attempt within 1 month prior to Week 0).
* Non-smoking subjects who self-reported "Never-Smoker" per the American Thoracic Society Questionnaire definition, and did not have urinary cotinine levels exceeding 50 ng/mL.
* Subjects, in the opinion of the Investigators, free of clinically significant health problems and not on medication on a daily basis for chronic medical disorders deemed clinically significant by the Investigator(s).
* Subjects not regularly taking creatine supplements.
* Subjects testing negative for selected drugs of abuse at Screening (included alcohol test).
* Subjects with a negative hepatitis panel (including hepatitis B surface antigen [HBsAg] and hepatitis C virus antibody [anti-HCV]) and negative Human Immunodeficiency Virus (HIV) antibody screens (for subjects immunized against hepatitis B with documentation of this immunization, a positive test result was not exclusionary).
* Female subjects who were non-pregnant (urine pregnancy test results were negative at Screening and Weeks 0, 12, and 24), non-lactating, and either postmenopausal (as verified by Follicle Stimulating Hormone levels) for at least 1 year, surgically sterile (e.g., tubal ligation, hysterectomy) for at least 90 days, or agreed to use from the time of signing the informed consent until 30 days after Week 24 (or Study Completion) a form of contraception considered acceptable to the Investigators (such as oral, injectable or implantable contraceptives, intrauterine devices and barrier methods ).
* Subjects able to read and comprehend questionnaires in English and willing to sign an Informed Consent Form.

Exclusion Criteria:

* Smokers using any other tobacco or nicotine-containing product or device other than tobacco-burning cigarettes from 6 months prior to the study through Week 24, including cigars, pipes, chewing tobacco, snuff, snus, nicotine patch, nicotine gum, etc.
* A history or clinical manifestations of significant metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, or psychiatric disorders.
* A history of hypersensitivity or allergies to any drug compound unless approved by the Investigator(s).
* A history or presence of an abnormal ECG deemed clinically significant by the Investigator.
* A history of alcoholism or drug addiction within 1 year prior to Study Entry.
* Evidence of visible oral cancer, as found in an oral health examination or based on oral health questions at each visit.
* Any acute or chronic condition that, in the Investigator(s)' opinion, limited the subject's ability to complete and/or participate in the study.
* Donation of blood from 30 days prior to Screening through Week 24 (or Study Completion), inclusive, or plasma from 2 weeks prior to Screening through Week 24 (or Study Completion), inclusive.
* Receipt of blood products within 2 months prior to Study Entry.
* Subject or a relative of the subject was currently or had ever been employed by the tobacco industry.
* Subject participated in any other investigational study drug or product trial in which receipt of an investigational study drug or product occurred within 30 days prior to Check-in (inclusive).

Ages: 28 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change in Urinary Tobacco Exposure Biomarkers from Weeks 0 to 12 | Week 12
  Nicotine and nine metabolites, tobacco-specific nitrosamines, polycyclic aromatic hydrocarbons, aromatic amines, benzene, isoprostanes, and urine mutagenicity
Change in Blood Tobacco Exposure Biomarkers from Weeks 0 to 12 | Week 12
  Lipid/cardiac risk markers, hypercoagulable state markers, endothelial function, DNA damage, and carboxyhemoglobin
Change in Markers of Exposure and Potential Harm from Weeks 0 to 12 | Week 12
  Exhaled carbon monoxide and spirometry
Change in health status scores from self-administered questionnaires on COPD-related disease from Weeks 0 to 12 | Week 12
  St. George's Respiratory Questionnaire and Leicester Cough Questionnaire
Change in tobacco usage diary from Weeks 0 to 4 | Week 4
Change in Urinary Tobacco Exposure Biomarkers from Weeks 0 to 24 | Week 24
  Nicotine and nine metabolites, tobacco-specific nitrosamines, polycyclic aromatic hydrocarbons, aromatic amines, benzene, isoprostanes, and urine mutagenicity
Change in Blood Tobacco Exposure Biomarkers from Weeks 0 to 24 | Week 24
  Lipid/cardiac risk markers, hypercoagulable state markers, endothelial function, DNA damage, and carboxyhemoglobin
Change in Markers of Exposure and Potential Harm from Weeks 0 to 24 | Week 24
  Exhaled carbon monoxide and spirometry
Change in daily tobacco usage diary from Weeks 4 to 8 | Week 8
Change in daily tobacco usage diary from Weeks 8 to 12 | Week 12
Change in daily tobacco usage diary from Weeks 12 to 16 | Week 16
Change in daily tobacco usage diary from Weeks 16 to 20 | Week 20
Change in daily tobacco usage diary from Weeks 20 to 24 | Week 24
Change in health status scores from self-administered questionnaires on COPD-related disease from Weeks 0 to 24 | Week 24
  St. George's Respiratory Questionnaire and Leicester Cough Questionnaire

SECONDARY OUTCOMES:
Change in Nicotine Yield versus Uptake from Weeks 0 to 12 | Week 12
  Mouth-level exposure to tar and nicotine
Change in health status scores from self-administered questionnaires on general health from Weeks 0 to 12 | Week 12
  Smoking Cessation Quality of Life Questionnaire (inclusive of the SF-36 v2)
Change in Nicotine Yield versus Uptake from Weeks 0 to 24 | Week 24
  Mouth-level exposure to tar and nicotine
Change in health status scores from self-administered questionnaires on general health from Weeks 0 to 24 | Week 24
  Smoking Cessation Quality of Life Questionnaire (inclusive of the SF-36 v2)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Ogden, Ph.D., Principal Investigator — R.J. Reynolds Tobacco Company
Locations (5):
- United States (5):
  - Covance Clinical Research Unit, Inc., Daytona Beach, Florida
  - Covance Clinical Research Unit, Inc., Boise, Idaho
  - Covance Clinical Research Unit, Inc., Portland, Oregon
  - Covance Clinical Research Unit, Inc., Austin, Texas
  - Covance Clinical Research Unit, Inc., Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogden MW, Marano KM, Jones BA, Stiles MF. Switching from usual brand cigarettes to a tobacco-heating cigarette or snus: Part 1. Study design and methodology. Biomarkers. 2015;20(6-7):382-90. doi: 10.3109/1354750X.2015.1094133. Epub 2015 Nov 2. PMID 26525849
- [Result] Ogden MW, Marano KM, Jones BA, Morgan WT, Stiles MF. Switching from usual brand cigarettes to a tobacco-heating cigarette or snus: Part 2. Biomarkers of exposure. Biomarkers. 2015;20(6-7):391-403. doi: 10.3109/1354750X.2015.1094134. Epub 2015 Nov 10. PMID 26554277
- [Result] Ogden MW, Marano KM, Jones BA, Morgan WT, Stiles MF. Switching from usual brand cigarettes to a tobacco-heating cigarette or snus: Part 3. Biomarkers of biological effect. Biomarkers. 2015;20(6-7):404-10. doi: 10.3109/1354750X.2015.1094135. Epub 2015 Nov 2. PMID 26525962